CLINICAL TRIAL: NCT05948280
Title: Virtual Reality-supported Mindfulness Practice in Relieving Stress in Postgraduate Students: a Pilot Randomised Controlled Trial
Brief Title: Virtual Reality (VR) Based Mindfulness Practice in Relieving Stress in Postgraduate Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Huiyuan LI, Postdoctoral Fellow, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CREC Ref. No. 2023.216
Record Dates: First submitted 2023-07-05; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Student; Stress; Virtual Reality; Mindfulness
Keywords: graduate student; stress; mental health; mindfulness; virtual reality
MeSH Terms: conditions — Psychological Well-Being | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Participants are assigned to three groups in parallel for the duration of the study. Participants in Group A receive Virtual reality-based mindfulness. Participants in Group B receive general mindfulness exercises. Participants in Group C receive no intervention as control.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor who is independent of the research will be trained before formally conducting data collecting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VR-supported mindfulness group (Experimental): Participants in the intervention group will receive VR mindfulness intervention, consisting of four face-to-face sessions (twice a week for two weeks). During the first week, the interventionist will teach and guide the participant face-to-face. During the second week, participants will be required to practice VR on their own for self-help.
  Interventions: Other: Virtual reality-supported mindfulness
- Mindfulness group (Active Comparator): Participants in this group will receive a mindfulness exercise guided by the interventionist twice a week for two weeks.
  Interventions: Other: Mindfulness
- Control group (No Intervention): Participants in the control group will not receive mindfulness or mindfulness plus VR.

INTERVENTIONS:
Other: Virtual reality-supported mindfulness — A single mindful stretching exercise provides a conscious stretch of VR scenario. The implementation of VR exercises will be performed by the interventionist who have received training in the application of VR scenarios and have extensive experience in VR research.
  Arms: VR-supported mindfulness group
Other: Mindfulness — The interventionist will guide the participant to do a mindful stretching exercise in the first week. During the second week, the interventionist will send participants an audio recording on how to do mindful stretching exercise via WeChat/WhatsApp.
  Arms: Mindfulness group

SUMMARY:
University students, especially graduate students, are constantly striving to achieve their goals, and their performance is constantly being evaluated, which creates a plethora of stressors, such as tests, a large amount of content to be learnt, lack of time, getting poor marks, and living up to their expectations. Mindfulness has been demonstrated to benefit one's emotions in a 'non-judgement' way. Evidence suggests that VR-based mindfulness practice may help individuals maintain present-moment awareness and block out distractions and may be more effective than conventional mindfulness approaches. The current pilot study aims to test the feasibility and acceptability of VR-based mindfulness practices in graduate students.

DETAILED DESCRIPTION:
A three-arm, assessor-blinded pilot randomised controlled trial (RCT) will be implemented. Participants will be randomly assigned to either mindfulness group, VR mindfulness group and control group. Participants will be randomised at a 1:1:1 ratio to the intervention groups or control group. Block randomization will be conducted by an independent research assistant using randomly varying block sizes of 4 and 6 to avoid selection bias. This study aims to test the feasibility, acceptability, and preliminary effects of the VR-based mindfulness practice in improving stress for graduate students.

Specific objectives are as follows:

1. To investigate the feasibility and acceptability of the VR-based mindfulness practice in improving stress for graduate students
2. To investigate the preliminary effects of VR-based mindfulness practice in improving stress for graduate students
3. To understand the user experience of mindfulness practice in VR

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 or over;
2. enrolled in graduate programme at the Chinese University of Hong Kong;
3. experienced stress: the score of perceived stress scale more than 13;
4. able to speak and write in English

Exclusion Criteria:

1. diagnosed with psychiatric disorders;
2. currently taking psychotropic medication;
3. have history of photosensitive epilepsy or previous experience of severe simulator sickness;
4. receiving or have just completed other psychological interventions (e.g. stress management, mental health support, peer support, etc) within the last six months will be excluded; or
5. history of seizures and motion sickness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Eligibility rate | Baseline
  The eligibility rate is defined as the percentage of participants fulfilling the inclusion criteria amongst the participants screened for the eligibility
Recruitment rate | Baseline
  The recruitment rate is defined as the percentage of participants who consented to participate in the study amongst the participants eligible for the study
Attrition rate | Week 2
  The attrition rate is defined as the percentage of participants who withdrew from the study before completion
Adherence rate | Week 2
  The adherence rate is defined as the frequency of the practice of mindfulness and session attendance
Change from baseline in the score of perceived stress assessed by The Perceived Stress Scale to immediately after the intervention | Baseline and Week 2 (post-intervention)
  A 10-item self-report instrument that measures the degree to which events are appraised as stressful and the frequency of perceived stressful situations. Students will be instructed to report the frequency of perceived stress over the past month from 0 (Never) to 4 (Very Often). Total scores on the PSS can range from 0 to 40. Higher total scores indicate higher levels of perceived stress.

SECONDARY OUTCOMES:
Change from baseline in the score of mindfulness assessed by The Five Facet Mindfulness Questionnaire to immediately after the intervention | Baseline and Week 2 (post-intervention)
  A 39-item self-report instrument that measures levels of mindfulness, including five facets: observing, describing, acting with awareness, non-judging of inner experience and non-reactivity to inner experience. Students will be invited to indicate on a 5-point Likert scale the degree to which each item is generally true for them, ranging from 1 to 5. Higher scores indicate higher levels of mindfulness.
Change from baseline in the level of mood states by The abbreviated Profile of Mood States to immediately after the intervention | Baseline and Week 2 (post-intervention)
  A 40-item self-report instrument that measures seven different subscales of transient mood states. Each question is score from 0 to 4. High scores indicate great mood disturbance.

OTHER OUTCOMES:
Acceptability of the intervention | Week 2
  Participants in the VR mindfulness group will be asked to provide qualitative feedback via a semi-structured interview. The interview questions focused on eliciting the participants' view about the VR experience, facilitators and barriers for VR-based mindfulness practice, and the positive and negative features of VR, which may help or hinder the mindfulness practice.

CONTACTS AND LOCATIONS:
Overall Officials: Cho Lee WONG, PhD, Study Director — The Nethersole School of Nursing, Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No